CLINICAL TRIAL: NCT01861041
Title: Low Dose, Low Concentration Different Baricity Bupivacaine for Transuretral Prostatectomy.
Brief Title: Low Dose Bupivacaine Spinal for Trans Uretral Prostatectomy.
Acronym: TURP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Reyhan Polat, Dr, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: PROSTAT
Record Dates: First submitted 2013-05-15; First posted 2013-05-23 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Benign Prostate Hyperplasia
Keywords: low dose; different baricity; spinal anesthesia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Heavy Bupivacain, Local anesthetic, Amp (Experimental): Heavy bupivacaine 7.5 mg (1.5 ml), 20 microgram fentanyl(0.4 ml), 1.1 ml saline , Total 3 ml
  Interventions: Drug: Heavy Bupivacaine
- Isobaric spinal, Local anesthetic, Amp (Active Comparator): 7,5 mg isobaric bupivacaine, 20 microgram (0.4 ml)fentanyl, 1.1 ml saline, Total 3 ml
  Interventions: Drug: Isobaric Bupivacaine

INTERVENTIONS:
Drug: Heavy Bupivacaine — 7,5 mg intrathecal hyperbaric bupivacain,
  Other Names: marcaine heavy
  Arms: Heavy Bupivacain, Local anesthetic, Amp
Drug: Isobaric Bupivacaine — 7.5 mg intratecal isobaric bupivacain
  Other Names: Marcain flakon
  Arms: Isobaric spinal, Local anesthetic, Amp

SUMMARY:
Spinal anesthesia, is used during the transuretheral resection of the prostate.Low dose hyperbaric local anesthetics have been used to enhance the resolution of the spinal block. We compared the efficacy and duration of the spinal block with two different bupivacaine baricities.

* Group I: low dose isobaric group
* GroupII: Low dose hyperbaric group

DETAILED DESCRIPTION:
Patients undergoing TURP were randomly allocated into two groups.

* Group I: Received fentanyl 20 µgr (0.4ml),heavy bupivacaine 0.5% (1.5 ml)and normal saline % 0.9 NaCl ( 1.1ml)
* Group II: Received fentanyl 20 µgr (0.4 ml), plain bupivacaine 0.5%(1.5 ml) normal saline 0.9% NaCl (1.1 mL) in total bupivacaine 0.25% (3ml) intrathecally.

Onset and duration of the sensory block, the degree of the motor block, side - effects and perioperative analgesic requirement assesed.

ELIGIBILITY:
Inclusion Criteria:

* 50-85 years ASA 1-4 BENİGN PROSTAT HYPERPLASİ

Exclusion Criteria:

* Allergy of study drugs
* Morbid obesity
* Spinal anesthesia contrindications
* Bleeding dyscrasias

Ages: 50 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2013-05; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Spinal Block Quality | 15 minute after intrathecal injection
  Sensory block assesment with pinpric test.

SECONDARY OUTCOMES:
Spinal block regression | 5 minute after arrival at PACU
  Sensory block assesment with pinprick test

CONTACTS AND LOCATIONS:
Overall Officials: MURAT M SAYIN, Ass. Prof, Study Director — Dispapi yildirim beyazit E R hospital
Locations (1):
- Diskapi Yildirim Beyazit Education and Research Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Loubert C, Hallworth S, Fernando R, Columb M, Patel N, Sarang K, Sodhi V. Does the baricity of bupivacaine influence intrathecal spread in the prolonged sitting position before elective cesarean delivery? A prospective randomized controlled study. Anesth Analg. 2011 Oct;113(4):811-7. doi: 10.1213/ANE.0b013e3182288bf2. Epub 2011 Sep 2. PMID 21890887
- [Background] Kim SY, Cho JE, Hong JY, Koo BN, Kim JM, Kil HK. Comparison of intrathecal fentanyl and sufentanil in low-dose dilute bupivacaine spinal anaesthesia for transurethral prostatectomy. Br J Anaesth. 2009 Nov;103(5):750-4. doi: 10.1093/bja/aep263. Epub 2009 Sep 28. PMID 19797249